CLINICAL TRIAL: NCT05968469
Title: The Effect of Aerobic Exercise Program on Disease Activity, Quality of Life, Spinal Mobility and Serum Calprotectin, Visfatin, Leptin,IL-33 Levels in Patients With Ankylosing Spondylitis: Ultrasonographic Study
Brief Title: The Effects of Aerobic Exercise in Patients With Ankylosing Spondylitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Afyonkarahisar Health Sciences University (Other)
Responsible Party: Principal Investigator, Faruk Emre Yulcu, Research Assistant Doctor, Physical Medicine and Rehabilitation, Afyonkarahisar Health Sciences University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ASHIIT2023
Record Dates: First submitted 2023-07-14; First posted 2023-08-01 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Ankylosing Spondylitis; Aerobic Exercise; Disease Activity
Keywords: Ankylosing Spondylitis; Spinal Mobility; Aerobic Exercise
MeSH Terms: conditions — Spondylitis, Ankylosing | interventions — Muscle Stretching Exercises

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Intensity Interval Training (HIIT) protocol (Experimental): Patients who underwent cycling ergometry program including high-intensity interval (HIIT) in the cardiopulmonary rehabilitation unit and stretching exercises for the cervical, thoracic and lumbar regions under the guidance of a physiotherapist
  Interventions: Device: Aerobic exercises with cycling ergometry
- Exercise program only: (Active Comparator): Patients undergoing cervical, thoracic and lumbar stretching exercises in the hospital with a physiotherapist
  Interventions: Other: Stretching exercises

INTERVENTIONS:
Device: Aerobic exercises with cycling ergometry — A total of 20 sessions of high-intensity interval (HIIT) aerobic exercise program will be applied to the patients using a bicycle ergometer, five days a week and once a day for four weeks. And then, it was planned to perform stretching exercises for the cervical, thoracic and lumbar regions and posture exercises accompanied by a specialist physiotherapist.
  The patients will be evaluated by the physician for a total of 3 times at the beginning of the treatment, at the end of the treatment (4th week) and at the 12th week after the start of the treatment. All patients will be evaluated for the parameters in the patient evaluation form, and blood samples taken between 08:00 and 10:00 in the morning and Calprotectin, Visfatin, Leptin, IL-33 serum levels will be measured with the ELISA kit.
  Arms: High Intensity Interval Training (HIIT) protocol
Other: Stretching exercises — Stretching exercises for the cervical, thoracic and lumbar regions and posture exercises were planned to be performed with the expert physiotherapist.
  The patients will be evaluated by the physician for a total of 3 times at the beginning of the treatment, at the end of the treatment (4th week) and at the 12th week after the start of the treatment. All patients will be evaluated for the parameters in the patient evaluation form, and blood samples taken between 08:00 and 10:00 in the morning and Calprotectin, Visfatin, Leptin, IL-33 serum levels will be measured with the ELISA kit.
  Arms: Exercise program only:

SUMMARY:
The aim of our study is to investigate the effects of aerobic exercise and stretching exercises applied in high-intensity interval training protocol on disease activity, quality of life, spinal mobility and calprotectin, visfatin, leptin, IL-33 serum levels in patients with Ankylosing Spondylitis.

DETAILED DESCRIPTION:
Ankylosing spondylitis (AS) is a painful and progressive chronic inflammation of the axial skeleton, mainly affecting the vertebral and sacroiliac joints. The management of AS aims to improve and maintain spinal mobility and normal posture, alleviate symptoms, reduce functional limitations and minimise complications. Due to the characteristic features of the disease, recommended spinal mobility exercises and aerobic exercises focus on reducing symptoms, improving functional capacity and quality of life, and improving and maintaining spinal mobility. Calprotectin, visfatin, leptin can be evaluated as biomarkers in inflammatory rheumatic diseases as an alternative to acute phase proteins and may reflect disease activity.

This study was designed as a prospective randomised controlled trial. Participants will be randomized into 2 groups and the intervention group will be given aerobic exercise and stretching exercise, and the other group only stretching exercise. BASDAI, BASMI, BASFI, ASQOL, ASDAS-CRP, Chest Expansion, 6 Minute Walk Test and Borg Scale will be used as assessment parameters.

Calprotectin, Visfatin, Leptin, IL-33 serum levels will be analysed by ELISA kit with blood samples taken in the early morning at the beginning of treatment, at the end of treatment (4th week) and at the 12th week after the beginning of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with ankylosing spondylitis according to 2009 ASAS diagnostic criteria,
* 20-60 years old, male and female gender,
* No change in anti-rheumatic drugs and dosage in the last 3 months
* Those who have not done regular physical activity in the last 3 months,
* Patients who do not have any orthopedic, neurological or mental illness that may affect exercise will be included in the study.

Exclusion Criteria:

* Active malignancy and/or history of malignancy in the last 5 years,
* Uncontrolled cardiopulmonary disease,
* Unstable angina pectoris, cardiac arrhythmias and myocardial infarction within the last 3 months
* Presence of pregnancy or those planning a pregnancy in the near future,
* History of major surgery (including joint surgery) within the last six months
* Use of assistive devices for ambulation or orthopaedic joint prosthesis
* Patients with total spinal ankyloses
* Patients with a history of syncope, exercise-induced arrhythmia
* Regular exercise in the last 3 months
* Patients with contracture of the knee joint that prevents cycling exercise

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2023-07-30 (Actual); Primary Completion 2024-10-21 (Actual); Study Completion 2025-01-12 (Actual)

PRIMARY OUTCOMES:
Change in BASDAI | Baseline, after 4 and 12 weeks
  The Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) consists of 6 questions about disease activity. Each question is scored on a scale of 0 to 10. High scores means high disease activity. It is a reliable and sensitive to changes index developed to assess disease activity and progression.

SECONDARY OUTCOMES:
Change in BASMI | Baseline, after 4 and 12 weeks
  The Bath Ankylosing Spondylitis Metrology Index (BASMI) is related to the spinal mobility of patients with ankylosing spondylitis. It consists of 5 clinical measurements. The total score of 5 measurements is obtained, the score range is between 0-10, a lower score means better spinal mobility.
Change in BASFI | Baseline, after 4 and 12 weeks
  The Bath Ankylosing Spondylitis Functional Index (BASFI) is a sensitive and reliable index developed for the determination and follow-up of functional status in patients with AS. It consists of 10 questions evaluating the functions of the patients. The final score is obtained by dividing the total score by 10 using the VAS in the range of 0-10 cm for each question. A high score indicates poor function.
Change in ASQOL | Baseline, after 4 and 12 weeks
  The Ankylosing Spondylitis Quality of Life Questionnaire (ASQoL) is the most widely used questionnaire to assess quality of life in AS, and it is valid and reliable. In this questionnaire consisting of eighteen questions, patients are asked to answer yes or no to each question. The total score varies between 0-18. High scores indicate serious deterioration in quality of life
Change in ASDAS-CRP | Baseline, after 4 and 12 weeks
  The Ankylosing Spondylitis Disease Activity Score-CRP (ASDAS-CRP) consists of four questions and the acute phase reactants CRP mg/L result. ASDAS-CRP will be calculated together with the CRP result in the formula. Mild disease activity <1.3 Moderate disease activity 1.3-2.1 High disease activity 2.1-3.5 Very high disease activity >3.5
Change in Chest Expansion | Baseline, after 4 and 12 weeks
  Chest expansion is determined by measuring the chest circumference following a deep inspiration and forced expiration. The expansion of the chest circumference is recorded in centimetres.
Change in 6 Minute Walk Test | Baseline, after 4 and 12 weeks
  The 6 Minute Walk Test is a sub-maximal exercise test used to assess aerobic capacity and endurance. The score of the test is the distance a patient walks in 6 minutes.
Change in Borg Scale | Baseline, after 4 and 12 weeks
  The Borg scale is a numerical expression of the verbal expression of exercise intensity in patients undergoing cycle ergometry. It allows direct comparison of individuals. 6 to 20 are evaluated. The Borg scale is a numerical expression of the verbal expression of exercise intensity in patients undergoing cycling ergometry. It allows direct comparison of individuals. 6 to 20 are evaluated. As the activity becomes more difficult for the patient, the values given increase.

CONTACTS AND LOCATIONS:
Overall Officials: Nuran EYVAZ, MD, Principal Investigator — Afyonkarahisar Health Sciences University
Locations (1):
- Afyonkarahisar Health Sciences University, Afyonkarahisar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yurdakul OV, Rezvani A. Can ultrasound be an assessment tool for sagittal spine mobility and chest expansion in patients with ankylosing spondylitis? Medicine (Baltimore). 2018 Sep;97(39):e12609. doi: 10.1097/MD.0000000000012609. PMID 30278577
- [Result] Jennings F, Oliveira HA, de Souza MC, Cruz Vda G, Natour J. Effects of Aerobic Training in Patients with Ankylosing Spondylitis. J Rheumatol. 2015 Dec;42(12):2347-53. doi: 10.3899/jrheum.150518. Epub 2015 Nov 1. PMID 26523029
- [Result] Diaconu AD, Ceasovschih A, Sorodoc V, Pomirleanu C, Lionte C, Sorodoc L, Ancuta C. Practical Significance of Biomarkers in Axial Spondyloarthritis: Updates on Diagnosis, Disease Activity, and Prognosis. Int J Mol Sci. 2022 Sep 30;23(19):11561. doi: 10.3390/ijms231911561. PMID 36232862
- See also: Can ultrasound be an assessment tool for sagittal spine mobility and chest expansion in patients with ankylosing spondylitis? — https://pubmed.ncbi.nlm.nih.gov/30278577/
- See also: Effects of Aerobic Training in Patients with Ankylosing Spondylitis — https://pubmed.ncbi.nlm.nih.gov/26523029/
- See also: Practical Significance of Biomarkers in Axial Spondyloarthritis: Updates on Diagnosis, Disease Activity, and Prognosis — https://pubmed.ncbi.nlm.nih.gov/36232862/